CLINICAL TRIAL: NCT04898257
Title: Effect of Lactibiane Tolerance®, a Multistrain Probiotic, to Treat Leaky Gut in Irritable Bowel Syndrome With Predominant Diarrhea (IBS-D) Patients: an Open-label, Single-center, Proof-of-concept, Pilot Study
Brief Title: Effect of Lactibiane Tolerance® to Treat Leaky Gut in Irritable Bowel Syndrome With Predominant Diarrhea (IBS-D)Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larena SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PILEJE-Lactibiane Tolerance
Record Dates: First submitted 2021-05-06; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This is a Phase IV, open-label, single-center, proof-of-concept, pilot study to evaluate the effect of Lactibiane Tolerance® in treating leaky gut in IBS-D patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactibiane Tolerance® (Other): 30 consecutive patients with IBS-D and an increased intestinal permeability assessed by 51Cr-EDTA or 99mTc-DTPA will receive the multistrain probiotic Lactibiane Tolerance® 10 billion CFU 1 capsule twice a day (30 minutes before breakfast and 30 minutes before dinner) for 30 days treatment. At the end of treatment, patients will repeat intestinal permeability assessment by 51Cr-EDTA or 99mTc-DTPA.
  Interventions: Dietary Supplement: Multistrain probiotic

INTERVENTIONS:
Dietary Supplement: Multistrain probiotic — After completion of screening phase, during baseline visit, eligible patients will be assigned to Lactibiane Tolerance® 10 billion CFU 1 capsule twice a day on an empty stomach (30 minutes before breakfast and 30 minutes before dinner).
  Other Names: Lactibiane Tolerance®

SUMMARY:
This is a Phase IV, open-label, single-center, proof-of-concept, pilot study to evaluate the effect of Lactibiane Tolerance® in treating leaky gut in IBS-D patients.

30 consecutive patients with IBS-D and an increased intestinal permeability assessed by 51Cr-EDTA or 99mTc-DTPA will receive the multistrain probiotic Lactibiane Tolerance® 10 billion CFU 1 capsule twice a day (30 minutes before breakfast and 30 minutes before dinner) for 30 days treatment. At the end of treatment, patients will repeat intestinal permeability assessment by 51Cr-EDTA or 99mTc-DTPA.

DETAILED DESCRIPTION:
Gut microbiota has many beneficial effects on the GI tract: barrier, immunomodulatory, metabolic, trophic among others. Microbiota unbalance or dysbiosis has been associated to digestive and extradigestive diseases.

Irritable bowel syndrome (IBS) is a common chronic disorder that affects the small and large intestine which causes cramping, abdominal pain, bloating, gas, diarrhea and/or constipation. Only a small number of people with IBS have severe signs and symptoms. Some people can control their symptoms by managing diet, lifestyle and stress. Others will need medication and counseling.

Intestinal permeability is the phenomenon of the gut wall in the gastrointestinal tract exhibiting permeability. It is a normal function of the intestine to exhibit some permeability, to allow nutrients to pass through the gut, while also maintaining a barrier function to keep potentially harmful substances (such as antigens) from leaving the intestine and migrating to the body more widely. In a healthy human intestine, small particles (< 4 Å in radius) can migrate through tight junction claudin pore pathways and particles up to 10-15 Å (3.5 kDa) can transit through the paracellular space uptake route. One way in which intestinal permeability is modulated is via CXCR3 receptors in the gut wall, which respond to zonulin. Gliadin (a glycoprotein present in wheat) activates zonulin signaling irrespective of the genetic expression of autoimmunity, leading to increased intestinal permeability to macromolecules. Bacterial pathogens such as cholera, select enteric viruses, and parasites modulate intestinal tight junction structure and function, and these effects may contribute to the development of chronic intestinal disorders. Excessive intestinal permeability is a factor in stress, infections and in some several autoimmune conditions such as Crohn's disease, celiac disease, type 1 diabetes, rheumatoid arthritis, spondyloarthropathies, inflammatory bowel disease and irritable bowel syndrome, but it is not clear if increased intestinal permeability is a cause or a consequence of these conditions.

According to its ability to modulate gut associated immune system, to compete with other GI bacteria and to increase enterocyte regeneration, probiotic therapy could be proposed to overcome an increased intestinal permeability. In particular, preliminary data suggested that the probiotic multistrains Lactibiane Tolerance® could be effective in Leaky gut treatment.

In fact, Nébot-Vivinus et al. demonstrated that Lactibiane Tolerance® could prevent epithelial barrier disruption induced by lipopolysaccharide, stress or colonic soluble factors from IBS patients and prevent visceral hypersensitivity in experimental models of epithelial barrier function.

Furthermore, Drouault-Holowacz et al. demonstrated that Lactibiane Tolerance® has anti-inflammatory properties in vitro by stimulating IL-10 production and in vivo by conferring a significant protective effect in the 2,4,6-trinitrobenzene sulfonic acid (TNBS)-induced colitis -induced colitis model (more than 50% decrease of colitis symptoms, P<0.01).This pilot study has been designed to evaluate the effect of multistrains probiotic Lactibiane Tolerance® in a consecutive subset of IBS-D patients with increased Intestinal permeability.

Subject participation in this study will be for approximately 45 days which includes up to a 2-week screening period and a 30-day treatment period.

All subjects will participate to the following visits: screening, enrolment, day 15 and day 30.

30 IBS-D patients Objectives Primary objective To demonstrate the effect of the multistrain probiotic Lactibiane Tolerance® in normalizing leaky gut in IBS-D patients Secondary objectives

* To characterize the effect of Lactibiane Tolerance® in improving symptoms of IBS
* To characterize the effect of Lactibiane Tolerance® on serum levels of zonulin
* To characterize the effect of Lactibiane Tolerance® on stool consistency
* To characterize the effect of Lactibiane Tolerance® on quality of life
* To evaluate the safety and tolerability of Lactibiane Tolerance®. Primary endpoint Proportion of subjects with normal intestinal permeability assessed by 51Cr-EDTA or 99mTc-DTPA after 30 days of treatment.

Secondary endpoints

* Mean variation of scores of items evaluated by VAS-IBS questionnaire after treatment compared to baseline
* Percentage of patients answering "yes" to the self-evaluation question: "Do you feel that your IBS symptoms have been satisfactory alleviated by this treatment?"
* Mean concentration of serum zonulin before and after treatment
* Mean score on Bristol Stool Scale before and after treatment and proportions of patients with 6 and 7 on Bristol Stool scale before and after treatment
* Mean score of IBSQoL questionnaire before and after treatment
* Safety and tolerability evaluated by the frequency of AEs, SAEs and AEs leading to discontinuation of study treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrolment into the study at baseline visit:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
2. Subjects are willing and able to participate in the study, complete subject assessments, attend scheduled clinic visits, and comply with all protocol requirements as evidenced by written informed consent.
3. Male and/or female subjects between the ages of ≥18 and ≤75 years at the time of informed consent.
4. Diagnosis of IBS following Rome IV criteria (Mearin et al., Gastroenterology 2016)*: Recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria:

   1. related with defecation
   2. associated with a change in frequency of stool
   3. onset associated with a change in form (appearance) of stool * Criteria fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.
5. Diagnosis of IBS with predominant diarrhea (IBS-D), following Rome IV criteria (Mearin et al., Gastroenterology 2016): more than one fourth (25%) of bowel movements with Bristol stool form types 6 or 7 and less than one-fourth (25%) of bowel movements with Bristol stool form types 1 or 2 or Patient reports that abnormal bowel movements are usually diarrhea (like type 6 or 7 in the picture of Bristol Stool Form Scale)
6. Evidence of a colonoscopy performed 5 years within the enrolment showing no evidence of organic disease
7. Evidence of increased intestinal permeability at 51Cr-EDTA or 99mTc-DTPA assessment performed during screening phase.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Subjects with suspect or evidence of organic disease, including but not limited to coeliac disease, inflammatory bowel disease, gastrointestinal neoplasia, unexplained anemia
2. Subjects with a history of colonic or small bowel resection.
3. Subjects with lactose intolerance
4. Use of probiotics or antibiotics or investigational agents within 30 days before baseline
5. Repeated use of anti-inflammatory drugs, including the non-steroidal anti-inflammatory drugs such as aspirin or ibuprofen within 7 days from the enrolment (except for prophylactic use of a stable dose of aspirin up to 325 mg / day for cardiac disease) and use of any product or ingredient that can have an effect on the intestinal permeability.
6. Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, immunologic, or local active infection/infectious illness) that, in the investigator's judgement will substantially increase the risk to the subject if he or she participates in the study.
7. Normal intestinal permeability at 51Cr-EDTA or 99mTc-DTPA assessment performed during screening
8. Women during pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with normal intestinal permeability assessed by 51Cr-EDTA or 99mTc-DTPA | 30 days
  To demonstrate the effect of the multistrain probiotic Lactibiane Tolerance® in normalizing leaky gut in IBS-D patients

SECONDARY OUTCOMES:
Mean variation of scores of items evaluated by VAS-IBS questionnaire after treatment compared to baseline | 30 days
  To characterize the effect of Lactibiane Tolerance® in improving symptoms of IBS.
Percentage of patients answering "yes" to the self-evaluation question: "Do you feel that your IBS symptoms have been satisfactory alleviated by this treatment?" | 30 days
  To characterize the effect of Lactibiane Tolerance® in improving symptoms of IBS.
Mean concentration of serum zonulin before and after treatment | 30 days
  To characterize the effect of Lactibiane Tolerance® on serum levels of zonulin
Mean score on Bristol Stool Scale before and after treatment | 30 days
  To characterize the effect of Lactibiane Tolerance® on stool consistency.
Proportions of patients with 6 and 7 on Bristol Stool scale before and after treatment | 30 days
  To characterize the effect of Lactibiane Tolerance® on stool consistency.
Mean score of IBSQoL questionnaire before and after treatment | 30 days
  To characterize the effect of Lactibiane Tolerance® on quality of life.
Safety and tolerability evaluated by the frequency of AEs, SAEs and AEs leading to discontinuation of study treatment. | 30 days
  To evaluate the safety and tolerability of Lactibiane Tolerance®.

CONTACTS AND LOCATIONS:
Overall Officials: Samira Aït Abdellah, Study Chair — Laboratoire PILEJE
Locations (1):
- Fondazione Policlinico Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No